CLINICAL TRIAL: NCT00969085
Title: Phase II Trial of Curcumin in Cutaneous T-cell Lymphoma Patients
Brief Title: Trial of Curcumin in Cutaneous T-cell Lymphoma Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0838
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Cutaneous T-cell lymphoma; Skin; Mycosis fungoides; MF; Sézary syndrome; SS; Curcumin; Turmeric
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Curcumin; Surveys and Questionnaires; Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curcumin (Experimental)
  Interventions: Drug: Curcumin (Turmeric); Behavioral: Questionnaires; Other: Photos

INTERVENTIONS:
Drug: Curcumin (Turmeric) — Chew then swallow 2 sticks per day for up to 6 months.
  2 sticks = 1 packet of curcumin = 8 grams
  Other Names: Turmeric
Behavioral: Questionnaires — Quality of life (QOL) questionnaires completed on Day 1, Weeks 2, 4, 8, 12, 16, 20, and at end of treatment visit.
  Other Names: Surveys
Other: Photos — Photos of up to 6 selected skin lesion(s) and half-body photos taken on Day 1, Weeks 2, 4, 12, and at end of treatment visit.
  Other Names: Pictures

SUMMARY:
The goal of this clinical research study is to learn if treatment with curcumin can help to decrease the size of lesions and/or decrease itching in patients with MF or SS. The safety of curcumin will also be studied.

DETAILED DESCRIPTION:
Curcumin:

Curcumin, a yellow substance taken from a plant, is commonly used in cooking as a spice called turmeric. In this study, participants will receive much higher doses of curcumin than can be received through food.

Curcumin may block proteins that help cells to divide. These proteins also may stop cancer cells from dying.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will swallow 2 sticks of curcumin per day. You should take the 2 sticks each morning with food and enough water for you to be able to swallow them. If you miss taking a dose of curcumin in the morning, you can take it later that day (as soon as you remember). However, if you miss a dose all day, do not take 2 doses the next day to make up for it.

Study Visits:

You will be asked to return for study visits.

At "baseline" (Day 1), the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked to rate your itching on a scale of 0-10.
* You will complete the 2 quality-of-life questionnaires.
* The study staff will take photos of up to 6 selected skin lesion(s). These will be close-up photos of the lesions and a small area of surrounding skin. "Half-body" photos will also be taken. These will be front, back, and/or side views of the top and bottom half of your body, depending on where the lesions are. For the half-body photos, your private areas will be covered (as much as possible), and your face will not be included in the photos unless there are lesions there.
* Blood (about 3 teaspoons) will be drawn for routine tests
* You will complete 2 "quality-of-life" questionnaires that ask how the symptoms of the disease may be affecting your life. This should take about 5 minutes.
* You will have a physical exam, including having skin lesions and affected areas of your skin looked at by the study doctor.
* If the study doctor thinks it is needed, you will have a skin biopsy performed. To perform a skin biopsy, the area is numbed with anesthetic and a small amount of tissue (about the size of a pencil eraser) is removed with a special tool.

The following tests and procedures will be performed at Weeks 2, 4, 8, 12, 16, and 20:

* You will have a physical exam, including having skin lesions and affected areas of your skin looked at by the study doctor.
* You will complete the 2 quality-of-life questionnaires.
* Your vital signs will be measured.
* You will be asked to rate your itching on a scale of 0-10.

At Weeks 2, 4, and 12 only, the following additional test will be performed:

-Just like at baseline, you will have skin lesion photos and half-body photos taken.

At Weeks 4, 12, and 20 only, the following additional test will be performed:

-Blood (about 3 teaspoons) will be drawn for routine tests.

If the doctor decides it is needed based on abnormal blood tests at screening, additional blood (about 1 teaspoon) will be drawn to check the status of the disease at Weeks 2, 4, 8, and 12.

If at any time during the study the skin disease seems to have cleared, you will have a skin biopsy performed in order to confirm the response.

Length of Study Participation:

You may continue receiving the study drug for up to 6 months, as long as you and the study doctor think you are benefitting from taking curcumin. If the disease gets worse or intolerable side effects occur at any time during this study, you will be taken off study.

End-of-Treatment Visit:

When you go off study for any reason, you will have an end-of-treatment visit. The following procedures will be performed:

* You will have a physical exam.
* You will be asked to rate your itching on a scale of 0-10.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor decides it is needed based on abnormal blood tests at screening, additional blood (about 1 teaspoon) will be drawn to check the status of the disease.
* A skin biopsy will be performed to check the status of the disease.
* Photos of the skin lesion(s) will be taken.
* You will complete the 2 quality-of-life questionnaires.
* You will have a CT and/or PET scan to check the size of the lymph nodes.

Follow-Up:

Every 3 months for 6 months after your last dose of the study drug, the study staff will check the results of any routine tests that were performed at your regular follow-up visits for MF or SS. If you do not visit the clinic during one or both of these two 3-month time periods, you will be called at home at 3 months and/or 6 months after your last dose of the study drug. The purpose of the phone calls is to ask how you are doing.

This is an investigational study. Curcumin is not FDA approved or commercially available for the treatment of cutaneous T-cell lymphoma. For this purpose, it is being used in research only.

Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has pathologically confirmed mycosis fungoides (MF) or Sézary syndrome (SS) form of cutaneous T-cell lymphoma (CTCL). Histology must be confirmed by the pathology department of the investigational center. This study is opened to MF and SS patients Stages 1A-IVA except for patients with aggressive disease requiring systemic chemotherapy. The patient must have pruritus at a severity of at least 3 to be eligible for the protocol.
2. The patient has been on a stable dose of antihistamine for at least two weeks and promises not to change the antihistamine or increase the dose.
3. The patient has a Karnofsky Performance Status of more than or equal to 60 at study entry.
4. The patient has given signed informed consent.
5. The patient has a life expectancy greater than 6 months.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count more than or equal to 1,500/mm^3, platelet count more than or equal to 100,000/mm^3.
7. The patient has adequate hepatic and renal function as defined by a total bilirubin less than or equal to 2.0 X ULN, alkaline phosphatase, AST and ALT less than or equal to 2.5 X ULN, and creatinine less than or equal to 2.0 mg/dL.
8. The patient agrees to practice effective contraception during the entire study period unless documentation of infertility exists. The methods of contraception include: abstinence, hormonal contraception (pills, injections, implants, and patches), intrauterine device, barrier methods (diaphragms, cervical caps, sponges, male and female condoms), and sterilization (vasectomy or tubal ligation). Women of childbearing potential are women who have not been menopausal for 12 consecutive months or have never been previously sterilized.
9. The patient is able to swallow curcumin powder.
10. The patient must also agree to refrain from use of additional herbal supplements.
11. There is no age limit for this protocol. Minor children will need to give assent with informed consent.

Exclusion Criteria:

1. The patient has a history of treated or active brain metastases, carcinomatous meningitis, an uncontrolled seizure disorder, or active neurological disease or has visceral disease stage IVB.
2. The patient has received prior local radiation treatment that would preclude evaluation for efficacy, or has received total body skin electron beam within 3 months prior to starting the trial.
3. The patient has an unstable medical condition according to the investigator, including, but are not limited to, an aggressive disease requiring systemic chemotherapy, uncontrolled diabetes mellitus Hgb A1c : >/= 8.or hypertension ( BP >/=140/90) or in the doctors opinion, active infections requiring systemic antibiotics, antivirals, or antifungals, unstable congestive heart failure, uncontrolled arrhythmias, unstable angina pectoris, unstable coagulation disorders, or psychiatric illness/social situations that would limit compliance with study requirements.
4. The patient is pregnant (confirmed by serum beta-HCG) or is breast feeding.
5. The patient is on any systemic therapy for MF/SS within the past 4 weeks, with the exception of Sézary syndrome patients, who may continue up to 10 mg of prednisone throughout trial participation.
6. The patient is on any topical therapy within the past 2 weeks, except if he/she has been using a stable dosage of topical steroids which does not exceed 2.5% hydrocortisone in MF patients, or triamcinolone 0.1% in Sézary syndrome patients. The patient must have been off high-potency steroids for at least 2 weeks. Moisturizers are allowed if they are not medicated and have been used for at least 2 weeks prior.
7. The patient has known HIV, active hepatitis B, and/or hepatitis C infection.
8. The patient currently has an active cancer other than CTCL that was diagnosed or had recurred in the last 2 years. The patient is allowed to participate if he/she has a history of skin cancers that have been treated.
9. The patient has known allergies to any component of the study drug.
10. The patient has any circumstances at the time of enrollment that would preclude completion of the study or the required follow-up.
11. The patient currently on active anticoagulation therapy (warfarin, aspirin, aspirin-containing products, NSAIDS or antiplatelet agents (eg, ticlopidine, clopidogrel, dipyridamole) who are at risk for platelet suppression.
12. The patient has biliary obstruction and/or elevated (greater than 2.5X normal) liver function studies (AST, ALT, and total bilirubin).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Response Rate using Physician's Global Assessment (PGA) based on Severity-Weighted Assessment Tool (SWAT) | Assessed every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org